CLINICAL TRIAL: NCT02217254
Title: A Prospective Multi-center Randomized Controlled Trial to Assess the Safety and Efficacy of One vs. Two Cryoablations Per Pulmonary Vein for the Treatment of Atrial Fibrillation
Brief Title: The OneFreeze Study
Acronym: OneFreeze
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UC-OF01
Record Dates: First submitted 2014-08-08; First posted 2014-08-15 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- two 3-minute cryoablations (Active Comparator): two 3-minute cryoablations per pulmonary vein during an atrial fibrillation ablation procedure
  Interventions: Procedure: Atrial fibrillation catheter ablation using the Medtronic Arctic Front Ablation System
- One 3-minute cryoablation (Active Comparator): One 3-minute cryoablation per pulmonary vein during an atrial fibrillation ablation procedure
  Interventions: Procedure: Atrial fibrillation catheter ablation using the Medtronic Arctic Front Ablation System

INTERVENTIONS:
Procedure: Atrial fibrillation catheter ablation using the Medtronic Arctic Front Ablation System
  Other Names: Pulmonary vein isolation; Cryoballoon catheter ablation

SUMMARY:
The One Freeze study is a prospective multi-center randomized controlled trial to assess the safety and efficacy of one vs. two cryoablations per pulmonary vein for the treatment of atrial fibrillation.

DETAILED DESCRIPTION:
The One Freeze Trial is an investigator-initiated trial that has been developed by the Principals at the University of California, San Francisco (UCSF) and with full participation of the Steering Committee. One Freezel is a prospective multicenter randomized controlled trial with a goal to enroll and randomize a minimum of 90 study participants. Participants will be randomized in a 1:1 ratio to either PVI with a single freeze per pulmonary vein (1F Group) or to PVI with at least two freezes per pulmonary vein (2F Group). The One Freeze study's primary aim is to determine if one 3-minute cryoablation per pulmonary vein results in a lower composite adverse event score as compared to the traditional method of using two 3-minute cryoablations per pulmonary vein.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation
* Age ≥ 18 years
* Life expectancy ≥ 1 year
* Willing and able to return to and comply with scheduled follow-up visits
* Willing and able to provide written informed consent

Exclusion Criteria:

* History of > 5 electric cardioversions
* History of previous pulmonary vein isolation ablation for atrial fibrillation
* History of MAZE procedure
* Left ventricular EF ≤ 35% within the past 12 months
* Mechanical mitral valve
* Single PV > 30 mm in diameter, unless deemed appropriate by the site PI
* Stroke/TIA within the past 6 months
* Creatinine > 2.0 mg/dL within the past 6 months
* Pregnancy or desire to get pregnant within the next 12 months
* Current enrollment in an investigation or study of a cardiovascular device or investigational drug that would interfere with this study
* Mental impairment or other conditions, which may not allow the participant to understand the nature, significance and scope of the study
* Any other condition or circumstance that in the judgment of the Clinical Site Investigator that makes the participant unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Composite Score of Adverse Events | 12 months
  Composite score of adverse events (Range 0-20 points) will be calculated after the patient has completed follow-up. Higher scores indicate greater severity.
  Luminal Esophageal Temperature (LET) (0-2 points): 1-point if ≤20 degrees C, 2-points if ≤15 degrees C
  Phrenic nerve injury (0-3 points): 1-point if ≥30% decrease in compound muscle action potential (CMAP) or loss of phrenic nerve capture resulting in cessation of freeze (without movement of pacing catheter), 2-points if Phrenic nerve palsy lasting> 1 minute resolving on table, 3-points if Phrenic nerve palsy not resolving on the table
  Pulmonary (0-4 points): 1-point if persistent dry cough > 1 week post ablation, 4-points if Hemoptysis
  Gastrointestinal (GI) (0-6 points): 1-point if Gastroparesis symptoms, 3-points if Esophageal ulceration, 6-points if left atrial-esophageal fistula
  Pulmonary vein (PV) stenosis (0-5 points): 1-point if ≥50% luminal area, 4-points if ≥90% luminal area, 5-points if total occlusion

SECONDARY OUTCOMES:
Participants free from symptomatic atrial fibrillation (AF) | 6 months and 12 months
  Participants experiencing no episodes of AF greater than 30 seconds, excluding episodes documented in the blanking period (6 weeks post-ablation for paroxysmal AF patients).
Atrial Fibrillation (AF) burden | 6 months, 12 months
  AF burden is defined as the overall percentage of AF during the 14-day observed period on Holter monitoring at 6 months and 12 months.
Procedure Time | 4 - 8 hours
  The duration of the Pulmonary Vein Isolation procedure from first leg puncture to removal of ablation catheter
Left Atrial Access time | 4 - 8 hours
  Time it takes to gain transseptal access during the catheter ablation procedure
Fluoroscopy Time | 4 - 8 hours
  The amount of time in minutes (and milligray (mGy)/millisievert (mSv) dosage) of fluoroscopy used during the procedure
Number of cryoablations needed to isolate each vein | 4 - 8 hours
  Number of cryoablations needed to isolate each vein
Acute success of the Pulmonary Vein Isolation (PVI) | 4 - 8 hours
  percentage of pulmonary veins isolated during the catheter ablation procedure
Individual Adverse Events | within 12 months after the Pulmonary Vein Isolation (PVI)
  Number and severity of adverse events following the PVI procedure during the 12-month follow-up window
Number of re-isolations required | 4 - 8 hours
  Number of pulmonary veins requiring touch up for re-isolation after initial isolation was achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Byron K Lee, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Virginia Mason Medical Center, Seattle, Washington
- Montreal Heart Institute, Québec, Canada